CLINICAL TRIAL: NCT02432924
Title: The Effect of Using Combined Personalised Instantaneous and Multidimensional Physical Activity Feedback on Motivation and Behaviour
Brief Title: Using Combined Instantaneous and Multidimensional Feedback to Support a Change in Physical Activity Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Max Western, Postgraduate researcher (PhD Candidate), University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EP-14/15-10
Record Dates: First submitted 2015-04-23; First posted 2015-05-04 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Motor Activity; Cardiovascular Diseases; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Motor Activity; Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback Group (Experimental): Participants randomised into the intervention group will be invited to return to the university for a one-off 60 minute set-up session once their physical activity monitor has been returned and processed. Within this session the participant will be given detailed instructions on how to use and wear the activity monitor and real time display and upload their data to and navigate the multidimensional feedback web platform (See materials section for details). They will also be introduced to the concept of goal setting and talked through the different aspects of the instantaneous feedback display and how that might benefit them. Following this visit the participant will be given licence to wear and use the physical activity monitoring devices for a 6-week period and encouraged to self-monitor their behaviour using the combined instantaneous and multidimensional feedback.
  Interventions: Behavioral: Instant + Multidimensional Physical Activity Feedback
- Waiting List Control Group (No Intervention): Participants who have been randomised into the control arm will be put on a 3 month waiting list to receive the intervention described above. They will still attend assessment visits at week 6 and week 12 while they are not receiving any advice or feedback. Following their 12 week assessment, participants in the control arm will be invited to attend the same 60 minute set-up session as received by the intervention group and then provided with the armband monitor and display to then receive the intervention in full. No further post-intervention or follow-up assessments will be taken from these participants.

INTERVENTIONS:
Behavioral: Instant + Multidimensional Physical Activity Feedback
  Other Names: Bodymedia
  Arms: Feedback Group

SUMMARY:
The primary aim of the study is to examine whether the provision of personalised multidimensional physical activity profiles (derived from technological advances in physical activity monitoring) is supported by instantaneous physical activity feedback in fostering a meaningful change in physical activity behaviour amongst adults.

DETAILED DESCRIPTION:
Advancements in monitoring technology not only permit the accurate capture of sophisticated physical activity information but also enable the provision of bespoke multidimensional feedback. Personalised feedback, self-monitoring and goal-setting are techniques that have been shown to be very effective in supporting a change in behaviour through improved motivation and awareness. To date the feedback provided in physical activity interventions invariably focuses on just one aspect of the behaviour and has had mixed results. Pedometers for example with a sole focus on the number of steps one takes has been shown to be a reasonably effective form of instant feedback in the short-term but its effects are rarely sustained after the device is removed. Tailored information about the achievement of 30 minutes of moderate to vigorous intensity activity is also only partially effective. One of the reasons might be that in focusing on just one aspect becomes prescriptive and doesn't allow individuals to explore the other important aspects that might be more aligned to their interests, needs and preferences. Having such narrow focused goals and information would likely frustrate rather than support an individual's needs for autonomy and competence, which is thought to be crucial in the adoption and maintenance of a new behaviour.

In this research, we want to find out whether the provision of both instantaneous and multidimensional personalised feedback about the different health-harnessing aspects of physical activity is effective in supporting adults in making a meaningful change to their physical activity behaviour. The study will take a mixed methods approach which will involve two phases. Phase 1 will involve a 2 group randomised control trial that will examine the use of combined instantaneous and multidimensional feedback over a 6-week period with a further follow-up outcome assessment a further 6-weeks after the intervention has finished. The second phase will involve a short one-to-one semi structured interview with each intervention participant that will be designed to qualitatively explore the preferred features of the intervention that were most effective for motivating and supporting a change in behaviour and/or to understand why it wasn't effective if applicable. The qualitative interviews will take place after the 6-week follow-up assessments have been completed so not to influence the results of any outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40-70 years inclusive
* Able to give informed consent to participate in the study

Exclusion Criteria:

* Diagnosed with coronary heart disease, chronic kidney disease (CKD stages 3-5), type 2 diabetes, stroke, heart failure and peripheral arterial disease
* Those with 'severe hypertension' defined as a BP greater than 180/110 mmHg.
* A BMI >40 kg/m2
* Use of weight loss drugs.
* A large recent (i.e. last 6 months) shift (>5%) in body mass or change in lifestyle.
* Those unable to change their physical activity (e.g. through disability or illness).
* Individuals who already lead highly physically active lifestyles (PAL > 2.0)
* Individuals who are not fluent in the English language.
* Pregnancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in physical activity level (PAL) | baseline, 6 weeks and 12 Weeks
  Mean physical activity level (PAL) as calculated using the formula average daily total energy expenditure/basal metabolic rate (Kcal). Minute by minute energy expenditure (TEE) will be objective measured using the SenseWear Armband (Bodymedia, software version 8.0). For assessment, monitors will be initialised with each individual's personal information (age, gender, height, and weight) and participants will be advised on how to fit and wear the devices. Participants will be asked to wear the monitor(s) for 7 days (including while sleeping) and will be asked to remove the monitors briefly for showers or water activities. As well as PAL the energy expenditure assessment will be used to determine total and average daily minutes of light intensity activity (greater than 1.5METs) moderate intensity activity (greater than 3METs); vigorous intensity activity (greater than 6 METs), accumulated moderate to vigorous activity bouts of 10 minutes and daily sedentary time.

SECONDARY OUTCOMES:
Motivation for Physical activity | baseline, 6 weeks and 12 Weeks
  Motivation for physical activity will be assessed using an adapted version of the behavioural regulations for exercise questionnaire (BREQ-2, Markland and Tobin, 2004).
Need satisfaction | baseline, 6 weeks and 12 Weeks
  Need satisfaction during physical activity will be measured by psychological need satisfaction in exercise (PNSE, Wilson et al., 2006).
Habitual physical activity | baseline, 6 weeks and 12 Weeks
  Habitual physical activity will be measured using the self-reported habit index (SRHI, Verplanken and Orbell, 2003).
Vitality | baseline, 6 weeks and 12 Weeks
  Vitality and quality of life will be assessed using the Subjective vitality index and Quality of life (SF-36, EQ-51) scales.
QIntervention: Change in cardiovascular disease and type 2 diabetes risk | baseline, 6 weeks and 12 Weeks
  Risk of Type 2 Diabetes and Cardiovascular disease will be calculated at http://qintervention.org/ and be ascertained from measurements of glucose and insulin control, C-Reactive Protein, fasting lipid profile (HDL:LDL ratio; total cholesterol and triglyceride) in the blood and height, weight, waist circumference, smoking status, blood pressure and familial history of CVD or diabetes. All of these measurements will be collected at the 3 assessment time points.

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Thompson, PhD, Study Director — University of Bath
Locations (1):
- University of Bath: Department for Health, Bath, United Kingdom

REFERENCES:
- [Derived] Western MJ, Standage M, Peacock OJ, Nightingale T, Thompson D. Supporting Behavior Change in Sedentary Adults via Real-time Multidimensional Physical Activity Feedback: Mixed Methods Randomized Controlled Trial. JMIR Form Res. 2022 Mar 2;6(3):e26525. doi: 10.2196/26525. PMID 35234658